CLINICAL TRIAL: NCT02179463
Title: A Multicenter Clinical Registry to Compare Different Patterns of Response Evaluation to Neoadjuvant Chemotherapy for Gastric Cancer
Brief Title: Compare Different Response Evaluations to Neoadjuvant Chemotherapy for Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jiafu Ji, Professor, Peking University
Other Study IDs: KW-NeoCT-Evaluation-2014; D141100000414004 (Other Grant/Funding Number: Beijing Municipal Science & Technology Commission)
Record Dates: First submitted 2014-06-21; First posted 2014-07-01 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Neoadjuvant chemotherapy; Response Evaluation
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Tumor, Blood Sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Neoadjuvant Chemotherapy: undergo neoadjuvant chemotherapy before surgery

SUMMARY:
RATIONALE: Neoadjuvant chemotherapy has been proved effective for locally advanced gastric cancer, yet the best pattern of response evaluation remain unknown.

PURPOSE: Compare different pattern of response evaluation for Gastric Cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Find the best pattern for response evaluation for gastric cancer. II. Assess the factor associated with this pattern.

OUTLINE: Neoadjuvant chemotherapy.

PROJECTED ACCRUAL: Up to 150 patients will be accrued over approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* sign written informed consent form
* age ≥ 18 years
* pathologically confirmed gastric or GEJ adenocarcinoma
* disease at clinical stage of locally advanced gastric cancer by CT/EUS(cT2+NanyM0)
* No prior antitumor treatment is allowed, including chemotherapy, radiotherapy, immune therapy or target therapy
* Adequate organ function as defined below:

Hematologic ANC ≥ 1.5*109/l Hemoglobin ≥ 9 g/dl Platelets ≥ 100*109/l Hepatic Albumin ≥ 30g/l Serum bilirubin ≤ 1.5×ULN AST and ALT ≤ 2.5×ULN ALP ≤ 2.5×ULN TBIL ≤ 1.5×ULN Renal Serum Creatinine < 1.5 ULN

* KPS ≥ 70
* Adequate lung and heart function
* Negative serum or urine pregnant test within 7 days prior to randomization for child-bearing age women
* Sexually active males or females willing to practice contraception during the study until 30 days after end of study.

Exclusion Criteria:

* Refuse to provide blood/tissue sample；
* With distant metastasis diagnosed by CT/EUS；
* Sexually active males or females refuse to practice contraception during the study until 30 days after end of study.
* History of organ transplantation（including autologous bone marrow transplantation and Peripheral stem cell transplantation）；
* Prior long term steroid therapy (excluding short term steroid treatment which is completed prior to > 2 weeks of study enrollment)；
* Patients with central nervous system(CNS) disorder or peripheral nervous system disorder or psychiatric disease；
* Concurrent severe infection；
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety (including current active hepatic, biliary, renal, respiratory disease, uncontrolled diabetes hypertension et al)；
* History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, are eligible；
* Known history of uncontrolled or symptomatic angina, uncontrolled arrhythmias and hypertension, or congestive heart failure, or cardiac infarction within 6 months prior to study enrollment, or cardiac insufficiency；
* Person with no capacity (legally) or inappropriate to continue study treatment for ethics/medical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced Gastric Cancer(cT2-4NanyM0)，estimated to do neoadjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pathological Response | 7days

SECONDARY OUTCOMES:
downstage proportion | 7days
  compared pathological stage with initial clinical stage, define T downstage or N downstage as downstage

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, MD, Principal Investigator — Peking University
Locations (1):
- Peking Unicersity Cancer Hospital, Beijing, Beijing Municipality, China